CLINICAL TRIAL: NCT00510835
Title: Protocolized Care for Early Septic Shock
Acronym: ProCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Derek C. Angus, MD, MPH, Chair, Critical Care Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P50GM076659 (NIH)
Record Dates: First submitted 2007-07-18; First posted 2007-08-02 (Estimated); Results first posted 2017-01-26 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2016-12

CONDITIONS: Sepsis; Severe Sepsis; Septic Shock
Keywords: septic shock; resuscitation; sepsis; cost-effectiveness; sepsis-induced organ dysfunction; early goal directed therapy; emergency medicine; critical care medicine
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Early Goal-Directed Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Early Goal Directed Therapy (EGDT) - The study team will insert a central venous catheter (CVC) for continuous monitoring of the subjects' central venous pressure (CVP) and central venous oxygen saturation (Scv02). The study team will use this information to give fluid, blood, and heart medications in a structured fashion. The CVC is FDA approved and routinely used in hospitals.
  Interventions: Procedure: Early Goal Directed Therapy (EGDT)
- 2 (Experimental): Protocolized Standard Care (PSC)- The study team will monitor the subjects' blood pressure and blood oxygen level with routine equipment. The study team will use this information to give fluid and heart medications in a structured fashion. CVCs will only be used when standard IVs are unable to give the proper amount of fluids and medicines. Blood transfusions will be given according to currently recommended guidelines.
  Interventions: Procedure: Protocolized Standard Care (PSC)
- 3 (Active Comparator): Usual Care - The attending physicians will treat the subjects according to their standard treatment plan and without any influence from the study team. A member of the study team will simply observe and record what happens.
  Interventions: Procedure: Usual Care (UC)

INTERVENTIONS:
Procedure: Early Goal Directed Therapy (EGDT) — Subjects will have a CVC inserted for continuous monitoring of their CVP and Scv02. Early structured treatment will be provided based on subjects' CVP, mean arterial pressure (MAP) and Scv02 measurements.
  Arms: 1
Procedure: Protocolized Standard Care (PSC) — Routine equipment will be used to monitor subjects' blood pressure and oxygen levels. Early structured treatment is based on the subjects' systolic blood pressure and the study doctors' judgment of fluid status and perfusion status.
  Arms: 2
Procedure: Usual Care (UC) — Attending physicians will provide routine care to subjects. Study measurements and treatments will be based on the physicians'/sites' standard practices.
  Arms: 3

SUMMARY:
The ProCESS study is large, 5-year, multicenter study of alternative resuscitation strategies for septic shock. The study hypothesizes that there are "golden hours" in the initial management of septic shock where prompt, rigorous, standardized care can improve clinical outcomes.

DETAILED DESCRIPTION:
Septic shock is a condition of acute organ dysfunction due to severe infection, with a mortality of up to 50%. Current efforts to improve care are limited by little practical evidence regarding the interventions in and timing of sepsis therapies. ProCESS is a prospective, randomized, three-arm parallel-group trial of alternative resuscitation strategies for early septic shock. The study objective is to improve the management of septic shock by exploring the clinical, biological, and economic aspects of alternative resuscitation strategies. This will be done by comparing two alternative resuscitation strategies to usual care in subjects with septic shock.

Comparisons:

1. Early Goal Directed Therapy (EGDT) - The subjects' blood pressure and blood oxygen levels will be monitored via the insertion of a central venous catheter (CVC). The study team will use this information to give fluid, blood and heart medications in a structured fashion. The central venous catheter to be used in this plan is FDA approved and routinely used in hospitals.
2. Protocolized Standard Care (PSC) - The subjects' blood pressure and blood oxygen levels will be monitored with standard equipment (without the CVC). The study team will use this information to prescribe fluid and heart medications in a structured fashion. CVCs will only be used when standard IVs cannot give the proper amount of fluids and medicines. Blood transfusions will be given according to currently recommended guidelines.
3. Usual Care (UC) - Subjects will be treated according to their attending physician's standard treatment plan and without any influence from the study team.

The primary hypotheses to be tested sequentially are that: protocolized resuscitation (EGDT and PSC) results in lower hospital mortality than usual care and Early Goal Directed Therapy results in lower hospital mortality than Protocolized Standard Care. These hypotheses will be tested on all enrolled subjects.

The study is powered to find an absolute mortality reduction (ARR) of ~6-7%. Based on the control arm mortality rate, we originally estimated a sample size of 1950. During the trial, the ProCESS Coordinating Center monitored the overall mortality rate, and appreciated that it was markedly lower than originally projected. Therefore, following a series of new calculations, in February 2013, the trial was re-sized to 1350 patients (450 patients per arm). The new size preserves the same power to find the same ARR. The resizing was fully blinded and approved by the NIH.

ELIGIBILITY:
Inclusion criteria:

* At least 18 years of age
* Suspected infection
* Two or more systemic inflammatory response syndrome (SIRS) criteria

  * Temperature </= 36˚ C or >/= 38˚C
  * Heart rate >/= 90 beats per minute
  * Mechanical ventilation for acute respiratory process or respiratory rate >/= 20 breaths per minute or PaC02 < 32 mmHg
  * WBC >/= 12,000/mm³ OR </= 4,000/mm³ OR > 10% bands
* Refractory hypotension (a systolic blood pressure < 90 mm Hg despite an IV fluid challenge of at least 1,000 mLs over a 30 minute period) or evidence of hypoperfusion (a blood lactate concentration >/= 4 mmol/L)

Exclusion criteria:

* Known pregnancy
* Primary diagnosis of acute cerebral vascular event, acute coronary syndrome, acute pulmonary edema, status asthmaticus, major cardiac arrhythmia, active gastrointestinal hemorrhage, seizure, drug overdose, burn or trauma
* Requirement for immediate surgery
* ANC < 500/mm³
* CD4 < 50/mm³
* Do-not-resuscitate status
* Advanced directives restricting implementation of the protocol
* Contraindication to central venous catheterization
* Contradiction to blood transfusion (e.g., Jehovah's Witness)
* Treating physician deems aggressive care unsuitable
* Participation in another interventional study
* Transferred from another in-hospital setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1351 (Actual)
Dates: Start 2008-03; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek C. Angus, MD, MPH, Principal Investigator — University of Pittsburgh; John A. Kellum, MD, Principal Investigator — University of Pittsburgh; Donald M. Yealy, MD, Principal Investigator — University of Pittsburgh
Locations (31):
- United States (31):
  - University of Alabama, Birmingham, Alabama
  - Maricopa Medical Center, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - LA County & USC Medical Center, Los Angeles, California
  - Stanford University School of Medicine, Palo Alto, California
  - UC Davis Medical Center, Sacramento, California
  - Norwalk Hospital, Norwalk, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Tampa General Hospital, Tampa, Florida
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Methodist Research Institute, Indianapolis, Indiana
  - Louisiana State University Health Sciences Center/Shreveport, Shreveport, Louisiana
  - University of Maryland/Baltimore, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - State University of New York - Downstate Medical Center, Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Summa Health System, Akron, Ohio
  - Penn State Hershey College of Medicine; Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Shadyside Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University Medical Center Brackenridge, Austin, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Intermountain Medical Center, Salt Lake City, Utah

REFERENCES:
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Background] Angus DC, Linde-Zwirble WT, Lidicker J, Clermont G, Carcillo J, Pinsky MR. Epidemiology of severe sepsis in the United States: analysis of incidence, outcome, and associated costs of care. Crit Care Med. 2001 Jul;29(7):1303-10. doi: 10.1097/00003246-200107000-00002. PMID 11445675
- [Background] Kochanek KD, Smith BL. Deaths: preliminary data for 2002. Natl Vital Stat Rep. 2004 Feb 11;52(13):1-47. PMID 14998175
- [Background] O'Brien PC, Fleming TR. A multiple testing procedure for clinical trials. Biometrics. 1979 Sep;35(3):549-56. PMID 497341
- [Background] Bone RC, Balk RA, Cerra FB, Dellinger RP, Fein AM, Knaus WA, Schein RM, Sibbald WJ. Definitions for sepsis and organ failure and guidelines for the use of innovative therapies in sepsis. The ACCP/SCCM Consensus Conference Committee. American College of Chest Physicians/Society of Critical Care Medicine. Chest. 1992 Jun;101(6):1644-55. doi: 10.1378/chest.101.6.1644. PMID 1303622
- [Background] Rivers EP, Ander DS, Powell D. Central venous oxygen saturation monitoring in the critically ill patient. Curr Opin Crit Care. 2001 Jun;7(3):204-11. doi: 10.1097/00075198-200106000-00011. PMID 11436529
- [Background] Feezor RJ, Baker HV, Mindrinos M, Hayden D, Tannahill CL, Brownstein BH, Fay A, MacMillan S, Laramie J, Xiao W, Moldawer LL, Cobb JP, Laudanski K, Miller-Graziano CL, Maier RV, Schoenfeld D, Davis RW, Tompkins RG; Inflammation and Host Response to Injury, Large-Scale Collaborative Research Program. Whole blood and leukocyte RNA isolation for gene expression analyses. Physiol Genomics. 2004 Nov 17;19(3):247-54. doi: 10.1152/physiolgenomics.00020.2004. PMID 15548831
- [Background] Maki DG, Stolz SM, Wheeler S, Mermel LA. Prevention of central venous catheter-related bloodstream infection by use of an antiseptic-impregnated catheter. A randomized, controlled trial. Ann Intern Med. 1997 Aug 15;127(4):257-66. doi: 10.7326/0003-4819-127-4-199708150-00001. PMID 9265424
- [Background] Pronovost P, Needham D, Berenholtz S, Sinopoli D, Chu H, Cosgrove S, Sexton B, Hyzy R, Welsh R, Roth G, Bander J, Kepros J, Goeschel C. An intervention to decrease catheter-related bloodstream infections in the ICU. N Engl J Med. 2006 Dec 28;355(26):2725-32. doi: 10.1056/NEJMoa061115. PMID 17192537
- [Background] McGee WT, Ackerman BL, Rouben LR, Prasad VM, Bandi V, Mallory DL. Accurate placement of central venous catheters: a prospective, randomized, multicenter trial. Crit Care Med. 1993 Aug;21(8):1118-23. doi: 10.1097/00003246-199308000-00008. PMID 8339574
- [Background] Goodnough LT, Brecher ME, Kanter MH, AuBuchon JP. Transfusion medicine. First of two parts--blood transfusion. N Engl J Med. 1999 Feb 11;340(6):438-47. doi: 10.1056/NEJM199902113400606. No abstract available. PMID 9971869
- [Background] Dodd RY, Notari EP 4th, Stramer SL. Current prevalence and incidence of infectious disease markers and estimated window-period risk in the American Red Cross blood donor population. Transfusion. 2002 Aug;42(8):975-9. doi: 10.1046/j.1537-2995.2002.00174.x. PMID 12385406
- [Background] Dellinger RP. Cardiovascular management of septic shock. Crit Care Med. 2003 Mar;31(3):946-55. doi: 10.1097/01.CCM.0000057403.73299.A6. No abstract available. PMID 12627010
- [Background] Hollenberg SM, Ahrens TS, Annane D, Astiz ME, Chalfin DB, Dasta JF, Heard SO, Martin C, Napolitano LM, Susla GM, Totaro R, Vincent JL, Zanotti-Cavazzoni S. Practice parameters for hemodynamic support of sepsis in adult patients: 2004 update. Crit Care Med. 2004 Sep;32(9):1928-48. doi: 10.1097/01.ccm.0000139761.05492.d6. PMID 15343024
- [Background] Rady MY, Smithline HA, Blake H, Nowak R, Rivers E. A comparison of the shock index and conventional vital signs to identify acute, critical illness in the emergency department. Ann Emerg Med. 1994 Oct;24(4):685-90. doi: 10.1016/s0196-0644(94)70279-9. PMID 8092595
- [Background] Yealy DM, Delbridge TR. The shock index: all that glitters.. Ann Emerg Med. 1994 Oct;24(4):714-5. No abstract available. PMID 8092601
- [Background] Rady MY, Rivers EP, Nowak RM. Resuscitation of the critically ill in the ED: responses of blood pressure, heart rate, shock index, central venous oxygen saturation, and lactate. Am J Emerg Med. 1996 Mar;14(2):218-25. doi: 10.1016/s0735-6757(96)90136-9. PMID 8924150
- [Derived] Fiorentino M, Xu Z, Smith A, Singbartl K, Palevsky PM, Chawla LS, Huang DT, Yealy DM, Angus DC, Kellum JA; ProCESS and ProGReSS-AKI Investigators. Serial Measurement of Cell-Cycle Arrest Biomarkers [TIMP-2] . [IGFBP7] and Risk for Progression to Death, Dialysis, or Severe Acute Kidney Injury in Patients with Septic Shock. Am J Respir Crit Care Med. 2020 Nov 1;202(9):1262-1270. doi: 10.1164/rccm.201906-1197OC. PMID 32584598
- [Derived] Massey MJ, Hou PC, Filbin M, Wang H, Ngo L, Huang DT, Aird WC, Novack V, Trzeciak S, Yealy DM, Kellum JA, Angus DC, Shapiro NI; ProCESS investigators. Microcirculatory perfusion disturbances in septic shock: results from the ProCESS trial. Crit Care. 2018 Nov 20;22(1):308. doi: 10.1186/s13054-018-2240-5. PMID 30458880
- [Derived] Hou PC, Filbin MR, Wang H, Ngo L, Huang DT, Aird WC, Yealy DM, Angus DC, Kellum JA, Shapiro NI; ProCESS Investigators( *). Endothelial Permeability and Hemostasis in Septic Shock: Results From the ProCESS Trial. Chest. 2017 Jul;152(1):22-31. doi: 10.1016/j.chest.2017.01.010. Epub 2017 Jan 19. PMID 28109962
- [Derived] ProCESS Investigators; Yealy DM, Kellum JA, Huang DT, Barnato AE, Weissfeld LA, Pike F, Terndrup T, Wang HE, Hou PC, LoVecchio F, Filbin MR, Shapiro NI, Angus DC. A randomized trial of protocol-based care for early septic shock. N Engl J Med. 2014 May 1;370(18):1683-93. doi: 10.1056/NEJMoa1401602. Epub 2014 Mar 18. PMID 24635773
- See also: ProCESS Study Web Site — https://crisma.upmc.com/processtrial/info2.asp

RESULTS

PARTICIPANT FLOW:
Groups:
- Early Goal Directed Therapy (EGDT): Early Goal Directed Therapy (EGDT) - The study team will insert a central venous catheter (CVC) for continuous monitoring of the subjects' central venous pressure (CVP) and central venous oxygen saturation (Scv02). The study team will use this information to give fluid, blood, and heart medications in a structured fashion. The CVC is FDA approved and routinely used in hospitals.
  Early Goal Directed Therapy (EGDT): Subjects will have a CVC inserted for continuous monitoring of their CVP and Scv02. Early structured treatment will be provided based on subjects' CVP, mean arterial pressure (MAP) and Scv02 measurements.
- Protocolized Standard Care (PSC): Protocolized Standard Care (PSC)- The study team will monitor the subjects' blood pressure and blood oxygen level with routine equipment. The study team will use this information to give fluid and heart medications in a structured fashion. CVCs will only be used when standard IVs are unable to give the proper amount of fluids and medicines. Blood transfusions will be given according to currently recommended guidelines.
  Protocolized Standard Care (PSC): Routine equipment will be used to monitor subjects' blood pressure and oxygen levels. Early structured treatment is based on the subjects' systolic blood pressure and the study doctors' judgment of fluid status and perfusion status.
- Usual Care: Usual Care - The attending physicians will treat the subjects according to their standard treatment plan and without any influence from the study team. A member of the study team will simply observe and record what happens.
  Usual Care (UC): Attending physicians will provide routine care to subjects. Study measurements and treatments will be based on the physicians'/sites' standard practices.
Period: Overall Study
Arm/Group | Early Goal Directed Therapy (EGDT) | Protocolized Standard Care (PSC) | Usual Care
Started | 445 | 448 | 458
Completed | 439 | 446 | 456
Not Completed | 6 | 2 | 2
Not completed — Withdrawal by Subject | 6 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Goal Directed Therapy (EGDT) | Protocolized Standard Care (PSC) | Usual Care | Total
Number analyzed (Participants) | 439 | 446 | 456 | 1341
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (16.4) | 61 (16.1) | 62 (16.0) | 61 (16.2)
Gender [Count of Participants; unit: Participants]
  Female | 207 | 194 | 192 | 593
  Male | 232 | 252 | 264 | 748
Region of Enrollment [Number; unit: participants]
  United States | 439 | 446 | 456 | 1341

OUTCOME MEASURES:

1. Primary Outcome: Hospital Mortality
Description: The primary study outcome is hospital mortality (defined as the number of deaths prior to discharge or 60 days, whichever comes first). The secondary outcomes are duration of survival (90 day and 1 year) and clinical evidence of organ dysfunction.
Time Frame: prior to discharge or 60 days, whichever comes first
Measure: Count of Participants; unit: Participants
Arm/Group | Early Goal Directed Therapy (EGDT) | Protocolized Standard Care (PSC) | Usual Care
Number analyzed (Participants) | 439 | 446 | 456
Participants | 92 | 81 | 86

2. Secondary Outcome: Changes in Markers of Inflammation, Oxidative Stress, Cellular Hypoxia and Coagulation/Thrombosis.
Time Frame: study hour 0, 6, 24 & 72
Reporting Status: Not Posted

3. Secondary Outcome: Resource Use and Costs of Alternative Resuscitation Strategies
Time Frame: at discharge or 60 days, whichever comes first
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were reported following the protocol guidelines: 1. Detailed information was collected regarding all SAEs that occurred during ProCESS study hours 0-72 2. Ongoing SAE information was collected for events related to the study PreSep line for the duration of the hospital stay or day 60 (whichever came 1st) 3. After hour 72, all SAEs that investigators considered potentially related to the study intervention were collected.
Arm/Group | Early Goal Directed Therapy (EGDT) | Protocolized Standard Care (PSC) | Usual Care
Serious Adverse Events (participants affected / at risk) | 23/439 | 22/446 | 37/456
Other Adverse Events (participants affected / at risk) | 41/439 | 49/446 | 52/456
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Early Goal Directed Therapy (EGDT) (N=439) | Protocolized Standard Care (PSC) (N=446) | Usual Care (N=456)
cardiac dysfunction (Cardiac disorders) | 7 | 5 | 7
gastrointestinal (Gastrointestinal disorders) | 0 | 0 | 2
hemorrhage/bleeding (Gastrointestinal disorders) | 0 | 0 | 1
hepatobiliary/pancreas (Hepatobiliary disorders) | 0 | 2 | 3
Infection (Infections and infestations) | 1 | 3 | 2
Metabolic/laboratory (Metabolism and nutrition disorders) | 2 | 3 | 3
neurology (Nervous system disorders) | 2 | 2 | 1
pain (General disorders) | 0 | 0 | 1 — Pain NOS
pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 10
renal/genitourinary (Renal and urinary disorders) | 5 | 1 | 5
vascular (Vascular disorders) | 1 | 1 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Early Goal Directed Therapy (EGDT) (N=439) | Protocolized Standard Care (PSC) (N=446) | Usual Care (N=456)
allergy/immunology (Immune system disorders) | 0 | 1 | 1
blood/bone marrow (Blood and lymphatic system disorders) | 5 | 7 | 8
cardiac dysfunction (Cardiac disorders) | 8 | 7 | 5
coagulation (Blood and lymphatic system disorders) | 2 | 2 | 0
dermatology/skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
endocrine (Endocrine disorders) | 0 | 0 | 1
gastrointestinal (Gastrointestinal disorders) | 3 | 2 | 3
hemorrhage/bleeding (Gastrointestinal disorders) | 0 | 1 | 1
hepatobiliary/pancreas (Hepatobiliary disorders) | 1 | 2 | 0
infection (Infections and infestations) | 1 | 3 | 3
lymphatics (Blood and lymphatic system disorders) | 0 | 0 | 1
metabolic/laboratory (Metabolism and nutrition disorders) | 3 | 8 | 14
neurology (Nervous system disorders) | 2 | 2 | 3
ocular/visual (Eye disorders) | 0 | 0 | 1
pain (General disorders) | 1 | 1 | 0
pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 9 | 11 | 3
renal/genitourinary (Renal and urinary disorders) | 2 | 2 | 1
vascular (Vascular disorders) | 3 | 0 | 5
hematoma (Surgical and medical procedures) | 0 | 0 | 1 — While remaining in the ICU, the subject developed a large hematoma in the right groin at the site of the femoral line and the line was removed. As this arm of the study is observational only this adverse event is considered unrelated to the study.
Line issue (Surgical and medical procedures) | 1 | 0 | 0 — Old line removed but unable to thread new line resulting in loss of CVL. Unable to access R IJ as shunt in place. Pt was to have central line surgically for hypotension, places upon admission to ICU and was determined not meet the criteria for SAE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No